CLINICAL TRIAL: NCT00490490
Title: Study of Bexxar <Tositumomab> Combined With External Beam Radiation Therapy for Patients With Relapsed, Bulky Non-Hodgkin's Lymphoma
Brief Title: Study of Bexxar <Tositumomab> Combined With External Beam Radiation Therapy
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Low Accrual
Sponsor: Stanford University (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Principal Investigator, Susan Knox, Associate Professor of Radiation Oncology, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-07479; 97437 (Other: Stanford University Alternate IRB Approval Number); LYMNHL0046 (Other: OnCore)
Record Dates: First submitted 2007-06-20; First posted 2007-06-22 (Estimated); Results first posted 2017-03-29 (Actual); Last update posted 2017-03-29 (Actual); Status verified 2017-02

CONDITIONS: Lymphoma, Non-Hodgkin
MeSH Terms: conditions — Lymphoma, Non-Hodgkin | interventions — tositumomab I-131; Radiotherapy; Potassium Iodide; Lugol's solution

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Tositumomab + XRT + KI (Experimental): Tositumomab + external beam radiotherapy (XRT) + potassium iodide (KI)
  Interventions: Drug: Bexxar (tositumomab); Procedure: External beam radiotherapy (XRT); Drug: Potassium Iodide (KI)

INTERVENTIONS:
Drug: Bexxar (tositumomab) — Tositumomab is a CD20-directed radiotherapeutic (131-iodine) monoclonal antibody indicated for the treatment of patients with CD20-positive, relapsed or refractory, low-grade, follicular, or transformed non-Hodgkin's lymphoma who have progressed during or after rituximab therapy, including patients with rituximab-refractory non-Hodgkin's lymphoma. Tositumomab (standard regimen) will be administered at whole body exposure of 75 cGy.
  Other Names: 131-iodine tositumomab
Procedure: External beam radiotherapy (XRT) — Patient-specific XRT will begin within 24 hours of administration of the therapeutic dose of tositumomab. Subjects will receive local XRT to bulky sites of disease measuring at least 5 cm in at least one dimension. The size and number of fields to be treated will determined by the investigators, but will encompass the patient's most symptomatic/threatening site(s) of disease and not cumulatively include more than 25% of the active bone marrow. Subjects will be treated with the 2 x 2 Gy regimen (2 daily fractions of 2 Gy). Sites of disease previously-irradiated with 30 to 40 Gy will not be treated on this study.
  Other Names: Radiotherapy (RT)
Drug: Potassium Iodide (KI) — Potassium iodide (KI) will be administered as:
  * Saturated solution potassium iodide (SSKI) 4 drops orally 3-times-a-day,
  * Lugol's solution 20 drops orally 3-times-a-day, OR
  * KI tablets 130 mg orally once per day KI treatment will start at least 24 hours prior to tositumomab, and continue daily for 14 days following the last dose of tositumomab
  Other Names: Saturated Solution Potassium Iodide (SSKI); Lugol's solution; Potassium iodide tablets

SUMMARY:
The purpose of the study is to assess the response rate of patients with relapsed or refractory low-grade or transformed low-grade, CD20-positive, B-cell non-Hodgkin's lymphoma to Iodine-131 (I-131) tositumomab (Bexxar) therapy plus local palliative radiation therapy (XRT).

DETAILED DESCRIPTION:
Response will be assessed on the basis of the presence or absence of measurable lesion ≥ 1.4 x 1.4 cm (operationally defined as ≥ 2.0 cm2) by radiographic evaluation OR ≥ 1.0 cm in greatest diameter detected by palpation on physical exam

ELIGIBILITY:
INCLUSION CRITERIA

* Histologically confirmed low grade CD20+ B cell non-Hodgkin lymphoma (NHL) patients who have relapsed after chemotherapy or are chemotherapy resistant and have one or more sites of disease measuring more than 5 cm.
* The patients must have failed at least one chemotherapy regimen
* No anticancer treatment for three weeks prior to study initiation (six weeks if Rituximab, nitrosourea or Mitomycin C)
* Fully recovered from all toxicities associated with prior surgery, radiation, chemotherapy or immunotherapy
* An institutional review board- (IRB)-approved signed informed consent
* Age 19 years or older
* Expected survival of at least 6 months
* Prestudy Performance Status of 0, 1 or 2 according to the World Health Organization (WHO)
* Absolute neutrophil count (ANC) of at least 1,500/mm³
* Platelet count at least 100,000/mm³
* Hct > 30%
* Hgb > 9.0 gm
* Bilirubin ≤ 2.0
* Creatinine ≤ 2.0
* Bone marrow involvement with lymphoma less than 25% (bilateral bone marrow) within 6 weeks of enrollment
* Acceptable birth control method for men and women

EXCLUSION CRITERIA

* Disease progression within 3 months of last chemotherapy
* Prior myeloablative therapies with bone marrow transplantation or peripheral stem cell rescue
* Platelet count less than 100,000/mm³
* Hypocellular bone marrow (≤ 15% cellularity)
* Marked reduction in bone marrow precursors of one or more cell lines
* History of failed stem cell collection
* Prior treatment with fludarabine
* Prior radioimmunotherapy
* Presence of central nervous system (CNS) lymphoma
* HIV or AIDS-related lymphoma
* Evidence of myelodysplasia on bone marrow biopsy
* Abnormal bone marrow cytogenetics
* Patients who have received prior external beam radiation therapy to more than 25% of active bone marrow
* Patients who have received filgrastim
* Sargramostim therapy within 3 weeks prior to treatment
* Presence of human anti-mouse antibody (HAMA) reactivity in patients with prior exposure to murine antibodies or proteins
* Serious nonmalignant disease or infection, which, in the opinion of the investigator and/or sponsor, would compromise other protocol objectives
* Another primary malignancy (other than squamous cell and basal cell cancer of the skin, in situ carcinoma of the cervix, or treated prostate cancer with stable prostate-specific antigen, PSA) for which the patients has not been disease free for at least 3 years
* Major surgery, other than diagnostic surgery within 4 weeks
* Pleural effusion
* Pregnant
* Lactating

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2007-01; Primary Completion 2011-06 (Actual); Study Completion 2013-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susan J Knox, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

RESULTS

PARTICIPANT FLOW:
Period: Completed Assessment for CR
Arm/Group | Tositumomab + XRT + KI
Started | 8
Completed | 8
Not Completed | 0
Period: Completed Assessment for TTP
Arm/Group | Tositumomab + XRT + KI
Started | 8
Completed | 5
Not Completed | 3
Not completed — Withdrawal by Subject | 1
Not completed — Lost to Follow-up | 2

BASELINE CHARACTERISTICS:
Arm/Group | Tositumomab + XRT + KI
Number analyzed (Participants) | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 5
  >=65 years | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 7
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 7
  More than one race | 0
  Unknown or Not Reported | 1
Histology [Count of Participants; unit: Participants] — Participants were staged according to the Ann Arbor Staging Classification System, as below.
  Stage / Characteristics
  1. Involvement of 1 lymphatic region
  2. Involvement of 2+ lymphatic regions on the same side of the diaphragm
  3. Involvement of lymphatic regions on both sides of the diaphragm
  4. Diffuse or disseminated involvement of 1+ extralymphatic organs
  Participants
    Follicular Lymphoma, Grade 1 | 2
    Follicular Lymphoma, Grade 2 | 2
    Follicular Lymphoma, Grade 3 | 2
    Marginal Zone B-Cell Lymphoma | 2

OUTCOME MEASURES:

1. Primary Outcome: Complete Response (CR) Rate
Description: Participants assessed for by the following Complete Response (CR) criteria
  CR or Functional CR
  * No evidence of disease and symptoms
  * Any macroscopic nodules detected in any organs no longer present.
  * Any palpable lymph node is normal and greatest diameter is < 1.0 cm.
  * The enlarged organs decreased in size and not palpable
  * The bone marrow biopsy and aspirate are negative for disease
  * Negative for disease by PET-scan (functional CR)
  CR Unconfirmed (CRu) criteria
  * No evidence of disease and symptoms
  * Any lymph node mass > 1.0 cm^2 diameter has regressed is size by more than 75%.
  * No macroscopic nodules in any organs
  * Any palpable lymph node is normal and greatest diameter is < 1.0 cm.
  * The bone marrow biopsy and aspirate are negative for disease
  * The bone marrow biopsy may have increased number or size of lymphoid aggregates without cytologic or architectural atypia
Time Frame: 12 weeks
Measure: Number; unit: percentage of participants
Arm/Group | Tositumomab + XRT + KI
Number analyzed (Participants) | 8
percentage of participants
  CR | 37.5
  Partial response (PR) or stable disease (SD) | 62.5

2. Secondary Outcome: Overall Response Rate (ORR)
Description: ORR is assessed as the sum of the overall rates of
  * CR confirmed by positron emission tomography (PET)
  * CR not confirmed by PET, and
  * Partial response (PR) negative for progression by PET
Time Frame: 12 weeks
Measure: Number; unit: percentage of participants
Arm/Group | Tositumomab + XRT + KI
Number analyzed (Participants) | 8
percentage of participants
  All CR + PR | 50
  Partial Response (PR) | 12.5
  Stable Disease (SD) | 50
  Progressive disease (PD) | 0

3. Secondary Outcome: Time-to-Progression (TTP)
Time Frame: 2 years
Population: One subject has not progressed (assessment not possible), and one subject has been lost to follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | Tositumomab + XRT + KI
Number analyzed (Participants) | 6
Participants
  3 months | 1
  6 months | 1
  9 months | 1
  18 months | 2
  60 months | 1

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | Tositumomab + XRT + KI
Serious Adverse Events (participants affected / at risk) | 8/8
Other Adverse Events (participants affected / at risk) | 8/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tositumomab + XRT + KI (N=8)
Anemia (Blood and lymphatic system disorders) | 3 (7)
Thrombocytopenia (Blood and lymphatic system disorders) | 8 (8)
Neutropenia (Blood and lymphatic system disorders) | 4 (10)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tositumomab + XRT + KI (N=8)
Anemia (Blood and lymphatic system disorders) | 8 (8)
Neutropenia (Blood and lymphatic system disorders) | 7 (7)
Thrombocytoperia (Blood and lymphatic system disorders) | 8 (8)
Back Pain (Musculoskeletal and connective tissue disorders) | 3 (3)
Body Aches (Musculoskeletal and connective tissue disorders) | 1 (1)
Bone Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 5 (5)
Leukocytopenia (Blood and lymphatic system disorders) | 8 (8)
Fatigue (General disorders) | 5 (14)
Burning sensation (Skin and subcutaneous tissue disorders) | 1 (1)
Chills (General disorders) | 1 (1) — Sweating, shock, shaking
Headaches (Nervous system disorders) | 8 (8)
Dizziness (Nervous system disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Equilibrium abnormal (Ear and labyrinth disorders) | 1 (1)
Body aches (General disorders) | 2 (2)
Infection, Finger (Infections and infestations) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Itchiness, hands and feet (Skin and subcutaneous tissue disorders) | 1 (1)
Mouth Sores (Infections and infestations) | 1 (3)
Neuropathy (Nervous system disorders) | 2 (2) — In fingers/toes
Skin Rash (Skin and subcutaneous tissue disorders) | 2 (2)
Sore Throat (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Stomach Pain (Gastrointestinal disorders) | 1 (1)
Swollem Lymph Nodes (Infections and infestations) | 1 (2) — L grion, R collarbone, L neck and back
Tremor (Nervous system disorders) | 1 (1)
Chest Pain (Cardiac disorders) | 1 (1)
Lung Infection (Infections and infestations) | 1 (1)
Indigestion (Metabolism and nutrition disorders) | 1 (1)
Back spasms (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in Hip/Leg (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain at biopsy site (lower back) (Musculoskeletal and connective tissue disorders) | 1 (1)
R Armpit Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain, side (Musculoskeletal and connective tissue disorders) | 1 (1) — Ribs hurt
Headache, Chronic (Nervous system disorders) | 1 (1)
Headaches (Nervous system disorders) | 5 (15)
Dizziness (Nervous system disorders) | 1 (2)
Itchiness, nose and mouth (Skin and subcutaneous tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No